CLINICAL TRIAL: NCT06277973
Title: Self-Care Immediate Stabilization Procedure (ISP) ® After a Traumatic Experience - A Feasibility Study
Brief Title: Feasibility Study of the Self-Care Immediate Stabilization Procedure (ISP) ® After a Traumatic Experience
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Oren Asman, Senior lecturer and director of the Samueli initiative for responsible AI in medicine, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0007551-2
Record Dates: First submitted 2024-02-11; First posted 2024-02-26 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Post-traumatic Stress Disorder; Acute Stress Disorder
Keywords: Post-traumatic stress disorder (PTSD); EMDR (Eye Movement Desensitization Reprocessing); Immediate Stabilization Procedure [IPS(R)]; The 'Butterfly Hug'; Acute Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic, Acute | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of the following groups: the experiment group and the waiting list group. Each group will receive the intervention but in the waiting list group this will occur a week later:
  Experiment group:
  Day 1 - questionnaires (T1) Day 4 - intervention Day 7 - questionnaires (T2) Day 97 - follow up questionnaires (T3)
  Waiting list group:
  Day 1 - questionnaires (T0) Day 7 - questionnaires (T1) Day 11- intervention Day 14- questionnaires (T2) Day 104- follow up questionnaires (T3) The parallel element of this model lies in the first week of the study: the experiment group goes through 2 measurements with the intervention in the middle of the week, whereas the waiting list group goes through 2 measurements without the intervention.
Who Masked: Participant
Masking Description: Participants will be informed that the intervention will occur between 2 days and 14 days and that they will fill 3-4 surveys. They will not be aware that there are two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Stabilization Procedure (Experimental): Participants in this arm will answer questionnaires and go through the intervention according to this schedule:
  Day 1 - questionnaires (T1) Day 4 - intervention Day 7 - questionnaires (T2) Day 97 - follow up questionnaires (T3)
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)
- Waiting list (Other): Participants in this arm will answer questionnaires and do the intervention according to this schedule:
  Day 1 - questionnaires (T0) Day 7 - questionnaires (T1) Day 11- intervention Day 14- questionnaires (T2) Day 104- follow up questionnaires (T3) Thus, unlike in the experimental arm, the intervention will be delayed by a week and participants will fill out questionnaires one additional time, a week before they begin the same protocol as the experimental arm.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — The intervention is based on EMDR therapy for PTSD treatment. Participants will answer demographic questions, choose a primary distress source and watch a therapist-guided video (male or female, based on participant choice) that will instruct them through the 'Butterfly Hug' method (tapping alternately on both sides of the body) while hearing positive statements from the therapists on the chosen distress source. Before and after each video participants will rate their distress level on a scale between 0 and 10 and they can view up to 8 videos per session. The system will monitor distress levels, and if it detects a sustained deterioration, it will end the intervention. At the end of the intervention, participants will be given information about possible reactions to it and how to deal with them, they will be encouraged to use the technique whenever necessary, and they will be informed of relevant support lines that they can contact if needed.

SUMMARY:
The study aims to assess the feasibility of an online intervention platform based on the Immediate Stabilization Procedure (ISP®). This intervention targets early trauma reactions, aiming to reduce the risk of future PTSD.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effectiveness and feasibility of an immediate stabilization procedure adapted for online self-usage.

This procedure relies on the Eye Movement Desensitization and Reprocessing (EMDR) treatment, a well-known approach for post-traumatic responses. It involves bilateral stimulation of the brain's hemispheres through tapping on the body (i.e., the 'Butterfly Hug') and positive therapist statements during the tapping process. Key advantages of this protocol include: 1) prevents long-term post-traumatic symptoms; 2) short intervention - takes 5-20 minutes on average; 3) simple procedure that does not require recalling traumatic memories; 4) could be administered by non-mental health experts.

The ISP® protocol was found effective and safe in Israel (face-to-face) and the Ukraine (remote). In addition, online variations of the protocol for self-usage have been utilized globally. The on-going state of war emphasizes the critical need for immediate emotional support. A collaborative group involving researchers, mental health clinicians, and software engineers adapted the ISP® protocol for online self-usage. The current study aims to evaluate the efficiency of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Hebrew speakers
2. Age 18 years or older
3. Have been in Israel since October 7th 2023 (the start of the war)
4. Were exposed to traumatic events during the war (Alarms, participated in battles, were attacked by terrorists, etcetera)
5. Access to PC/smartphone
6. Basic technological skills, ability to use the internet and email.

Exclusion Criteria:

1. Diagnosed with psychotic conditions.
2. Diagnosed with PTSD or complex PTSD.
3. Diagnosed with alcohol use disorder or drug abuse disorder.
4. Suicidal ideation
5. Treated with medication, psychotherapy, or any other mental treatment

About 10 randomly selected subjects will perform the intervention while recorded via zoom in the presence of a research assistant. This will allow us to assess the way subjects utilize this intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
PCL-5 (Posttraumatic Stress Disorder Checklist) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The PCL-5 is a self-report 20-item questionnaire that conforms with the DSM-5 symptom criteria for PTSD. Each item is rated on a scale of 0-4 and reflects a symptom of PTSD and the total scores range from 0 to 80. The severity scores for DSM-5 symptom clusters can be obtained by adding the scores for the items within each cluster, i.e., cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20).
GAD-7 (General Anxiety Disorder-7) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  A widely used self-report measure for assessing symptoms of generalized anxiety disorder is the Generalized Anxiety Disorder-7 (GAD-7). Moreover, it can also be used to measure anxiety in the general population. This questionnaire contains seven items, and the final questionnaire result is the sum of the items. The total score ranges from 0 to 21, with each item's scale ranging from 0 to 3.
  0-4: minimal anxiety 5-9: mild anxiety 10-14: moderate anxiety 15-21: Severe anxiety
SSASI (The Short Scale Anxiety Sensitivity Index) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The Short Scale Anxiety Sensitivity Index (SSASI) is a shorter version of the Anxiety Sensitivity Index-3 (ASI-3).
  This 5-items scale measures an individual's fear of the negative consequences associated with anxiety symptoms (i.e. anxiety sensitivity). Each item's scale ranges from 0 (very little) to 4 (very much).
BSI 18 (Brief Symptom Inventory) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The Brief Symptom Inventory-18 (BSI-18) is a self-report measure consisting of 18 items, designed to effectively assess general mental health. Each item represents a symptom, and respondents are asked to rate these symptoms on a five-point scale, based on how much they have been bothered by the symptom in the prior week. The BSI-18 measure has three dimensions: somatization, depression, and anxiety; each contains 6 items.
DES-II (Dissociative Experiences Scale) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The DES-II is a self-administered 28-item questionnaire, designed to measure the frequency of dissociative experiences of individuals. Score in this questionnaire ranges from 0 to 100, with higher score indicating higher dissociative symptoms and severity. For each item, respondents indicate how often a particular experience occurred to them, from "never" (0% of the time) to "always" (100%).
DERS (Difficulties in Emotion Regulation Scale) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) is a self-report measure that assesses individuals' typical levels of difficulties in emotion regulation. The total score ranges from 16 to 80, with higher scores indicating greater difficulty regulating emotions.
NSESSS (The National Stressful Events Survey Acute Stress Disorder Short Scale) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The National Stressful Events Survey Acute Stress Disorder Short Scale (NSESSS) is a 7-item scale that assesses the severity of acute stress disorder symptoms after experiencing a highly stressful event or experience. Each item is rated on a 5-point scale, with 0 indicating 'Not at all' and 4 indicating ' Extremely'. Individuals are asked to rate the severity of his or her posttraumatic stress disorder during the past 7 days. The total score can range from 0 to 28, with higher scores indicating greater severity of acute stress disorder.
SASRQ (Stanford Acute Stress Reaction Questionnaire) | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  The SASRQ is a 30-item self-report questionnaire that is designed to evaluate the severity of traumatic stress symptoms over the past four weeks. The total score in this measure ranges from 0 to 150, with higher scores indicating more severe traumatic stress symptoms.
Exposure to traumatic event during the current war | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  This measure will be composed of 4 items that will require participants to indicate whether they have experienced a traumatic event during the current war. Participants will need to specify the type of traumatic event, its severity and whether they have begun a psychological/ psychiatric treatment during this time.
  In the first baseline session the questions will refer to exposure to traumatic events during the war (up to the present moment). In all subsequent sessions, exposure to traumatic events will refer to events that occurred since the latest session.
PDEQ (Peritraumatic Dissociative Experiences Questionnaire) | Experimental group - day 1, waiting list group - days 1 and 7
  The PDEQ is a self-report questionnaire consisting of 10 items, designed to assess peritraumatic dissociation. Respondents are asked to rate on a 5-point Likert scale ranging from 1 (Not at all true) to 5 (Extremely true), based on how much each statement relates to their experience during the traumatic event. The PDEQ has well-established psychometric properties, with higher total scores indicating increased peritraumatic dissociation.
TIS (Tonic Immobility Scale) | Experimental group - day 1, waiting list group - days 1 and 7
  TIS is a commonly used questionnaire to assess tonic immobility during traumatic events. This self-report instrument is divided into two parts: Tonic Immobility (7 items) and Fear (3 items). Each item is rated on a 7-point Likert scale. The range of the total score is between 0 and 60, with higher scores indicating more tonic immobility and fear during the event.
PDI (The Peritraumatic Distress Inventory) | Experimental group - day 1, waiting list group - days 1 and 7
  The PDI questionnaire is used to measure distress at the time of injury and consists of 13 items, with responses given on a 4-point Likert scale. The total score can range from 0 to 52, with higher scores representing greater symptom burden.
Questionnaires to test user experience of the system | Experimental group - day 7, waiting list group - day 14
  This questionnaire will be composed of 7 items on a 7-point scale and is designed to evaluate the system's ease of use, the degree to which it is easy to learn it, and its overall user experience. Higher total scores will represent a more positive user experience from the system.
Questionnaire for examining the experience of the intervention | Experimental group - day 7, waiting list group - day 14
  This questionnaire will consist of 3 items on a 7-point scale and will be used to assess the participant's satisfaction with the intervention, the extent to which it is helpful, and the overall experience. Higher total scores will represent a more positive user experience from the system.
Qualitative interview | Experimental group - day 97, waiting list group - day 104
  Approximately 20 subjects from the original sample will participate in a qualitative interview that will last about 30 minutes. The questions of the interview will focus on the experience of the participant from the system and their thought on its content.
Questionnaire regarding receiving emotional treatment | Experimental group - days 1, 7 and 97. Waiting list group - days 1, 7, 14 and 107
  Participants will be asked whether they have received emotional treatment (psychological, counseling, etc.) or medication since entering the study.

CONTACTS AND LOCATIONS:
Overall Officials: Oren Asman, LLD, Principal Investigator — Tel Aviv University; Yael Lahav, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available (upon request) to other researchers. potentially identifying information will be removed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It will be available after completion of the study and with the submission of research articles based on it for review and publication (estimation - May 2025)
Access Criteria: Academic researchers focusing on mental trauma and or digital wellbeing interventions.

REFERENCES:
- [Background] Beatty, S., Moore-Felton, M.S., Zaporozhets, O. et al. Effectiveness of Immediate Stabilization Procedure (ISP®) Associated with Wartime Events. Int J Adv Counselling (2023). https://doi.org/10.1007/s10447-023-09531-2
- [Background] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Background] Brunet A, Weiss DS, Metzler TJ, Best SR, Neylan TC, Rogers C, Fagan J, Marmar CR. The Peritraumatic Distress Inventory: a proposed measure of PTSD criterion A2. Am J Psychiatry. 2001 Sep;158(9):1480-5. doi: 10.1176/appi.ajp.158.9.1480. PMID 11532735
- [Background] Cardena E, Koopman C, Classen C, Waelde LC, Spiegel D. Psychometric properties of the Stanford Acute Stress Reaction Questionnaire (SASRQ): a valid and reliable measure of acute stress. J Trauma Stress. 2000 Oct;13(4):719-34. doi: 10.1023/A:1007822603186. PMID 11109242
- [Background] Derogatis LR. BSI 18, Brief Symptom Inventory 18: Administration, scoring and Procedure Manual. Minneapolis, MN: NCS Pearson, Incorporated; 2001.
- [Background] Fuse T, Forsyth JP, Marx B, Gallup GG, Weaver S. Factor structure of the Tonic Immobility Scale in female sexual assault survivors: an exploratory and Confirmatory Factor Analysis. J Anxiety Disord. 2007;21(3):265-83. doi: 10.1016/j.janxdis.2006.05.004. Epub 2006 Jul 18. PMID 16854560
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Kilpatrick DG, Resnick HS, Milanak ME, Miller MW, Keyes KM, Friedman MJ. National estimates of exposure to traumatic events and PTSD prevalence using DSM-IV and DSM-5 criteria. J Trauma Stress. 2013 Oct;26(5):537-47. doi: 10.1002/jts.21848. PMID 24151000
- [Background] Marmar, C. R., Weiss, D. S., & Metzler, T. J. (1997). The Peritraumatic Dissociative Experiences Questionnaire. In J. P. Wilson & T. M. Keane (Eds.), Assessing psychological trauma and PTSD (pp. 412-428). The Guilford Press.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 10(4), 206
- [Background] Zvolensky MJ, Garey L, Fergus TA, Gallagher MW, Viana AG, Shepherd JM, Mayorga NA, Kelley LP, Griggs JO, Schmidt NB. Refinement of anxiety sensitivity measurement: The Short Scale Anxiety Sensitivity Index (SSASI). Psychiatry Res. 2018 Nov;269:549-557. doi: 10.1016/j.psychres.2018.08.115. Epub 2018 Aug 29. PMID 30199696